CLINICAL TRIAL: NCT05473182
Title: IndieTrainer: Enabling Individuals With Cerebral Palsy to Receive Gamified Power Mobility Training in Their Own Manual Wheelchairs
Brief Title: IndieTrainer: Enabling Individuals With Cerebral Palsy to Receive Power Mobility Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Principal Investigator, Lisa Kenyon, Professor, Grand Valley State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-278-H
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Conditions Similar to Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: One group pretest-posttest design with a single session retention trial 4 weeks after the end of the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: All child participants receive the intervention (Other): All child participants receive power wheelchair skills training using the IndieTrainer system.
  Interventions: Other: IndieTrainer system

INTERVENTIONS:
Other: IndieTrainer system — The IndieTrainer system is comprised of the IndieGo device and video-game modules. The IndieGo device temporarily converts a manual wheelchair into a powered wheelchair, thereby allowing children to remain in their own manual wheelchair and use their own custom seating system during power wheelchair skills training activities. The video-game modules are integrated into the IndieGo device such that the video games can be played on a TV screen using the specific access method used to control the IndieGo (i.e., switch or joystick). The IndieTrainer system is designed to allow a child to practice power wheelchair skills as part of the video-game modules or as part of more traditional power wheelchair skills training activities wherein children are able to actively explore the environment and practice executing actual wheelchair skills.

SUMMARY:
Power wheelchairs offer children who are unable to independently opportunities for participation in social, educational, and leisure activities. Unfortunately, children who have severe cognitive, motor, or sensory impairments may need extended training to be able to master the power wheelchairs skills needed to "qualify" for their own power wheelchairs. The IndieTrainer system was developed to address this need. The IndieTrainer system is comprised of the IndieGo device and video-game modules. The IndieGo device temporarily converts a manual wheelchair into a powered wheelchair, thereby allowing children to remain in their own manual wheelchair and use their own custom seating system during power wheelchair skills training activities. The video-game modules are integrated into the IndieGo device such that the video games can be played on a television screen using the specific access method used to control the IndieGo (i.e., switch or joystick). The IndieTrainer system is designed to allow a child to practice power wheelchair skills as part of the video-game modules or as part of more traditional power wheelchair skills training activities wherein children are able to actively explore the environment and practice executing actual wheelchair skills. This study will evaluate the use of the IndieTrainer system in children with cerebral palsy, ages 3-21 years.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of cerebral palsy or similar conditions with functional abilities consistent with a Gross Motor Classification System Classification System Level IV or Level V
* Inability to functionally self-propel a manual wheelchair
* Does not have an individually prescribed powered wheelchair
* Currently using a manual wheelchair or adaptive stroller that can be safely used with the IndieTrainer system (i.e., functioning wheel brakes to remain locked onto platform, etc.) as assessed by the PI
* Has at least one parent/caregiver who is able to converse in English (as assessed by the PI during interactions over the phone and in person) due to safety concerns

Exclusion Criteria:

* Any condition or issue that would prevent a child from safely using the IndieTrainer system as determined by the PI, a licensed physical therapist.
* The child and his/her manual wheelchair or adaptive stroller combined must weigh <300 pounds to safely use the IndieTrainer.

  * A diagnosis of a progressive condition with the potential for functional decline across the study period, such as spinal muscular atrophy, Duchenne muscular dystrophy, etc.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Consist with NIH requirements, at the conclusion of the study, deidentified data collected in this study will be placed in a repository where it can be accessed by other researchers for future studies.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD will be made available 6 months following publication of study results
Access Criteria: Study results and summaries will be publicly available at clinicaltrials.gov. For specific IPD, the study PI and co-investigators will review all requests for data sharing. Data will be shared for purposes of secondary analysis, contribution to a population-related database, or similar reasons that are intended to advance the evidence-based provision of family-centered care for children with disabilities.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although child-parent/caregiver dyads were enrolled in this study, only child participants received the intervention.
Period: Overall Study
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Started | 25 (Child/parent or caregivers dyads were enrolled in this study. The enrollment number provided represents the number of dyads (25 children and 25 parents/caregivers). Note: Only child participants received the intervention.)
Completed | 25 (Child/parent or caregivers dyads were enrolled in this study. The enrollment number provided represents the number of dyads (25 children and 25 parents/caregivers). Note: Only child participants received the intervention.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for parents/caregivers.
Groups:
- Single Arm: All Child Participants Receive the Intervention: All child participants receive power wheelchair skills training using the IndieTrainer system.
  IndieTrainer system: The IndieTrainer system is comprised of the IndieGo device and video-game modules. The IndieGo device temporarily converts a manual wheelchair into a powered wheelchair, thereby allowing children to remain in their own manual wheelchair and use their own custom seating system during power wheelchair skills training activities. The video-game modules are integrated into the IndieGo device such that the video games can be played on a TV screen using the specific access method used to control the IndieGo (i.e., switch or joystick). The IndieTrainer system is designed to allow a child to practice power wheelchair skills as part of the video-game modules or as part of more traditional power wheelchair skills training activities wherein children are able to actively explore the environment and practice executing actual wheelchair skills. Baseline data were not collected for parents/caregivers.
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Months] | 109 (47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Assessment of Learning Powered Mobility Use [Mean (Standard Deviation); unit: units on a scale] | 2.24 (.78)

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Participants' Understanding How to Use a Power Mobility Device Between Baseline and Immediately After the Conclusion of the Intervention Period at Week 3
Description: This outcome will be assessed using each child participant's score (from a minimum of 1 to a maximal of 8) on the Assessment of Learning Powered mobility use. The Assessment of Learning Powered mobility use measures a child's understanding of how to use a power mobility device. Higher scores indicate a better outcome.
Time Frame: From baseline to immediately after the conclusion of the intervention period at Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 2.68 (0.8524)

2. Primary Outcome: Change in Child Participants' Power Mobility Skill Performance Between Baseline and Immediately After the Conclusion of the Intervention Period at Week 3
Description: This outcome will be assessed using the Wheelchair Skills Checklist that evaluates a child's performance of 7 items, each reflecting a specific power mobility skill. Each item is scored from a minimum of 0 to a maximum of 2 with a higher score indicating a better outcome. Total scores for all 7 items range from a minimum of 0 to a maximum of 14 with higher scores therefore indicate a better outcome.
Time Frame: From baseline to immediately after the conclusion of the intervention period at Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 1.1486 (0.3535)

3. Primary Outcome: Change in Parental/Caregiver Perceptions of Their Child's Power Mobility Skills Performance Between Baseline and Immediately Following the End of the Intervention Period at Week 3.
Description: This outcome will be assessed using the Canadian Occupational Performance Measure to rate parent/caregiver perceptions of their child's performance of 5 power mobility skills. Each skill is rated from a minimum of 1 to a maximum of 10. A higher score indicates a better outcome. The total score on all 5 items ranges from a minimum of 5 to a maximum of 50. A higher score indicates a better outcome.
Time Frame: From baseline to immediately after the conclusion of the intervention period at Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 6.864 (1.4739)

4. Primary Outcome: Change in Child Participants' Understanding How to Use a Power Mobility Device From Immediately After the Conclusion of the Intervention Period at Week 3 to the End of the Follow-up Period at Week 7
Description: as for outcome 1
Time Frame: From immediately after the conclusion of the intervention period at Week 3 to the end of the follow-up period at Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 0.16 (0.3742)

5. Secondary Outcome: Parent/Caregiver Satisfaction With the IndieTrainer System Intervention Immediately After the Conclusion of the Intervention at Week 3
Description: This outcome will be assessed through use of the Client Satisfaction Questionnaire-8 an 8-item questionnaire exploring stakeholder satisfaction with an intervention. Response choices for each item range from minimum of 1 to a maximum of 4. Higher scores indicate higher satisfaction. Total scores on the Client Satisfaction Questionnaire-8 range from a minimum of 8 to a maximum of 32. Higher total scores indicate higher satisfaction with the intervention.
Time Frame: Immediately after the conclusion of the intervention at Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 31.52 (.77)

6. Primary Outcome: Change in Child Participants' Power Mobility Skill Performance Between the Conclusion of the Intervention Period at Week 3 and the End of the Follow up Period at Week 7.
Description: as for outcome 2
Time Frame: From immediately after the conclusion of the intervention period at Week 3 to the end of the follow-up period at Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm: All Child Participants Receive the Intervention
Number analyzed (Participants) | 25
score on a scale | 0.0514 (0.0911)

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Adverse event data were only collected for child participants. Adverse event data were not collected for parents/caregivers.
Groups:
- Single Arm: All Participants Receive the Intervention: All participants receive power wheelchair skills training using the IndieTrainer system.
  IndieTrainer system: The IndieTrainer system is comprised of the IndieGo device and video-game modules. The IndieGo device temporarily converts a manual wheelchair into a powered wheelchair, thereby allowing children to remain in their own manual wheelchair and use their own custom seating system during power wheelchair skills training activities. The video-game modules are integrated into the IndieGo device such that the video games can be played on a TV screen using the specific access method used to control the IndieGo (i.e., switch or joystick). The IndieTrainer system is designed to allow a child to practice power wheelchair skills as part of the video-game modules or as part of more traditional power wheelchair skills training activities wherein children are able to actively explore the environment and practice executing actual wheelchair skills.
Arm/Group | Single Arm: All Participants Receive the Intervention
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05473182/Prot_SAP_000.pdf